CLINICAL TRIAL: NCT05304611
Title: Safety and Efficacy of L9LS, a Human Monoclonal Antibody Against Plasmodium Falciparum, in a Dose-Escalation Trial in Adults and Children and a Randomized, Double-Blind Trial of Children in Mali
Brief Title: Anti-malaria MAb in Malian Children
Acronym: L9LS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH); Malaria Research and Training Center, Bamako, Mali (Other); University of the Sciences, Techniques and Technologies of Bamako (Other); University of Washington (Other); Harvard School of Public Health (HSPH) (Other); Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022/34/CE/USTTB
Record Dates: First submitted 2022-02-28; First posted 2022-03-31 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Plasmodium Falciparum Infection; Malaria
MeSH Terms: conditions — Malaria | interventions — Injections, Subcutaneous; Injections, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Adult Dose-escalation study: Arm 1: 300 mg of L9LS (Experimental): Adult participants receive single dose of 300 mg of L9LS subcutaneously. Once subjects reach day 7 post-administration without safety concerns dosing begins for arm 2.
  Interventions: Biological: L9LS (VRC-MALMAB0114-00-AB) Subcutaneous injection
- Adult Dose-escalation study: Arm 2: 600 mg of L9LS (Experimental): Adult participants receive single dose of 600 mg of L9LS subcutaneously. Once subjects reach day 7 post-administration without safety concerns dosing begins for arm 3.
  Interventions: Biological: L9LS (VRC-MALMAB0114-00-AB) Subcutaneous injection
- Adult Dose-escalation study: Arm 3: 20 mg/kg of L9LS (Experimental): Adult participants receive highest single dose of 20 mg/kg IV of L9LS intravenously. Once subjects reach day 7 post-administration without safety concerns dosing begins for pediatric subjects dose escalation arm 1.
  Interventions: Biological: L9LS (VRC-MALMAB0114-00-AB) intravenous injection
- Pediatric Dose-escalation study: Arm 1: 150 mg of L9LS (Experimental): Pediatric subjects ages 6-10 years receive single dose of 150 mg L9LS subcutaneously. Once subjects reach day 7 post-administration without safety concerns, dosing begins for arm 2.
  Interventions: Biological: L9LS (VRC-MALMAB0114-00-AB) Subcutaneous injection
- Pediatric Dose-escalation study: Arm 2: 300 mg of L9LS (Experimental): Pediatric subjects ages 6-10 years receive single dose of 300 mg L9LS subcutaneously. Once subjects reach day 7 post-administration without safety concerns, dosing begins for the pediatric efficacy study arms.
  Interventions: Biological: L9LS (VRC-MALMAB0114-00-AB) Subcutaneous injection
- Pediatric Dose-escalation study: Arm 3: Placebo (Placebo Comparator): Pediatric subjects ages 6-10 receive single dose placebo of normal saline subcutaneously for comparison.
  Interventions: Other: Placebo
- Pediatric Efficacy study: Arm 1: 150 mg of L9LS (Experimental): Pediatric subjects ages 6-10 receive single dose of 150 mg L9LS subcutaneously.
  Interventions: Biological: L9LS (VRC-MALMAB0114-00-AB) Subcutaneous injection
- Pediatric Efficacy study: Arm 2: 300 mg of L9LS (Experimental): Pediatric subjects ages 6-10 receive single dose of 300 mg L9LS subcutaneously.
  Interventions: Biological: L9LS (VRC-MALMAB0114-00-AB) Subcutaneous injection
- Pediatric Efficacy study: Arm 3: Placebo (Placebo Comparator): Pediatric subjects ages 6-10 receive single dose placebo of normal saline subcutaneously.
  Interventions: Other: Placebo
- Pediatric Extension study: Arm 1: 150 mg of L9LS (Experimental): Pediatric subjects ages 6-10 who completed year one of the study and agreed to continue with the extension were randomized to receive 150 mg of L9LS subcutaneously.
  Interventions: Biological: L9LS (VRC-MALMAB0114-00-AB) Subcutaneous injection
- Pediatric Extension study: Arm 2: 300 mg of L9LS (Experimental): Pediatric subjects ages 6-10 who completed year one of the study and agreed to continue with the extension were randomized to receive 300 mg of L9LS subcutaneously.
  Interventions: Biological: L9LS (VRC-MALMAB0114-00-AB) Subcutaneous injection
- Pediatric Extension study: Arm 3: Placebo (Placebo Comparator): Pediatric subjects ages 6-10 who completed year one of the study and agreed to continue with the extension were randomized to receive placebo of normal saline subcutaneously.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: L9LS (VRC-MALMAB0114-00-AB) Subcutaneous injection — Administered one time via subcutaneous route.
  Arms: Adult Dose-escalation study: Arm 1: 300 mg of L9LS; Adult Dose-escalation study: Arm 2: 600 mg of L9LS; Pediatric Dose-escalation study: Arm 1: 150 mg of L9LS; Pediatric Dose-escalation study: Arm 2: 300 mg of L9LS; Pediatric Efficacy study: Arm 1: 150 mg of L9LS; Pediatric Efficacy study: Arm 2: 300 mg of L9LS; Pediatric Extension study: Arm 1: 150 mg of L9LS; Pediatric Extension study: Arm 2: 300 mg of L9LS
Biological: L9LS (VRC-MALMAB0114-00-AB) intravenous injection — Administered one time via intravenous route.
  Arms: Adult Dose-escalation study: Arm 3: 20 mg/kg of L9LS
Other: Placebo — Normal saline administered one time via subcutaneous route.
  Arms: Pediatric Dose-escalation study: Arm 3: Placebo; Pediatric Efficacy study: Arm 3: Placebo; Pediatric Extension study: Arm 3: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of onetime subcutaneous (SC) or intravenous (IV) administration of monoclonal antibody (MAb) L9LS in healthy Malian adults and one-time SC administration of L9LS in healthy Malian children, as well as its protective efficacy against naturally occurring Plasmodium falciparum (Pf) infection over a 7-month malaria season in healthy Malian children 6-10 years of age.

DETAILED DESCRIPTION:
A two-part, phase 2 trial evaluating the safety and tolerability of onetime subcutaneous (SC) or intravenous (IV) administration of monoclonal antibody (MAb) L9LS in healthy Malian adults and one-time SC administration of L9LS in healthy Malian children, as well as its protective efficacy against naturally occurring Plasmodium falciparum (Pf) infection over a 7-month malaria season in healthy Malian children 6-10 years of age.

The first part of the study is an age de-escalation and dose-escalation study for safety and tolerability. Adult subjects in the dose-escalation study will be assigned in open-label fashion to 1 of 3 L9LS dose arms. Dosing will begin in the lowest dose arm. Once all subjects in that arm reach day 7 post-administration, if no safety concerns have arisen, dosing will begin at the next dose level. Once all subjects in that arm reach day 7 post-administration, if no safety concerns have arisen, dosing will begin at the highest dose level. Once all adult subjects reach day 7 post-administration, if no safety concerns have arisen, 18 subjects aged 6-10 years will be randomized 1:1 to L9LS or placebo in double-blind fashion. Once all 18 subjects reach day 7 post-administration, if no safety concerns have arisen, an additional 18 subjects aged 6-10 years will be randomized 1:1 to L9LS versus placebo. Randomization of subjects aged 6-10 years in each L9LS dose arm will be weight-stratified and enrollment will be weight de-escalated. Adult subjects will be followed for safety to assess adverse events (AEs) at study visits 1, 3, 7, 14, 21, and 28 days after administration, and once every month thereafter through 28 weeks. Subjects aged 6-10 years will be followed at study visits 1, 3, 7, 14, 21, and 28 days after administration, and once every 2 weeks thereafter through 36 weeks. Primary study assessments include physical examination and blood collection for identification of Pf infection and other research laboratory evaluations. After the last subject in the pediatric L9LS dose arm reaches day 7 safety follow-up, an interim safety evaluation will be performed before enrollment begins for the efficacy part of the study. Data from the 36 subjects aged 6-10 years enrolled in the dose-escalation study will be included in a secondary analysis to determine the relationship between L9LS concentration and the risk of Pf infection.

The second part of the study is a weight-stratified, randomized, double-blind, placebo-controlled trial to assess safety and protective efficacy of L9LS versus placebo administered SC in children 6-10 years of age. In this part of the study, subjects will be randomized to L9LS or placebo. Randomization of subjects in each arm will be weight-stratified. Subjects in the efficacy study will receive the study agent prior to the malaria season and be followed at study visits 1, 3, 7, 14, 21, and 28 days later, and once every 2 weeks thereafter through 24 weeks. Primary study assessments include physical examination and blood collection for identification of Pf infection and other research laboratory evaluations.

Prior to the last study visit of the original protocol described above (January 2023 - February 2023), study participants who remain enrolled in the dose-escalation and efficacy studies will be invited to participate in a 12-month extension study. After the safety and efficacy results are unblinded (approximately March/April 2023), participants who agree to continue with the extension will be grouped into one of 3 arms based on their original study arm assignment:

Arm 1: Up to 84 subjects who received 150 mg of L9LS in year 1 (9 from the dose-escalation study, plus 75 from the efficacy study).

Arm 2: Up to 84 subjects who received 300 mg of L9LS in year 1 (9 from the dose-escalation study, plus 75 from the efficacy study).

Arm 3: Up to 93 subjects who received placebo in year 1 (18 from the dose-escalation study, plus 75 from the efficacy study).

The protocol extension employs a pre-specified, adaptive design based on the time-to-event efficacy of 150 mg and 300 mg of L9LS against P. falciparum infection as detected by blood smear observed after the first malaria season in the original protocol. Specifically, if 150 mg and 300 mg of L9LS both show ≥60% efficacy during the first malaria season (based on the upper bound of the two-sided 95% confidence interval [CI]), participants will be re-randomized 1:1 in a double-blind fashion within each arm to receive a single dose of either L9LS (150 or 300 mg depending on study arm) or placebo administered SC before the 2023 malaria season.

The same randomization scheme will be followed if in the first malaria season the 300-mg dose of L9LS shows ≥60% efficacy (based on the upper bound of the two-sided 95% CI) and the 150-mg dose of L9LS shows <60% efficacy (based on the upper bound of the two-sided 95% CI) but the difference between their respective point estimates of efficacy is ≤10%, with the exception that children who received placebo in year 1 will receive 300 mg of L9LS (or placebo) in year 2.

If 300 mg of L9LS shows ≥60% efficacy (based on the upper bound of the two-sided 95% CI) and 150 mg of L9LS shows <60% efficacy (based on the upper bound of the two-sided 95% CI) but the difference between their respective point estimates of efficacy is >10% during the first malaria season, participants will be re-randomized 1:1 in a double-blind fashion within each arm to receive a single dose of either 300 mg of L9LS or placebo administered SC before the 2023 malaria season.

If 150 mg and 300 mg of L9LS both show <60% efficacy (based on the upper bound of the two-sided 95% CI) after the first malaria season, the protocol extension will be abandoned.

Before study agent administration, all subjects will be given artemether-lumefantrine to clear any preexisting Pf blood-stage infection.

Subjects will be followed at study visits 1, 3, 7, 14, 21, and 28 days after administration, and once every 2 weeks thereafter through 28 weeks, with a final visit occurring on study day 252 (36 weeks) to collect a final PK sample. Primary study assessments include medical history, physical examination, and blood collection for pharmacokinetics (PK), anti-drug antibody (ADA) assessments, identification of Pf infection by microscopic examination of thick blood smears and RT-PCR, and other research laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Is within the appropriate age range for the respective cohort:

  1. Children: Aged ≥6 years and <11 years.
  2. Adults: Aged ≥18 years.
* Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
* In good general health and without clinically significant medical history.
* Adult participants or parent and/or guardian of minor participants able to provide informed consent.
* Willing to have blood samples and data stored for future research.
* Resides in or near Kalifabougou or Torodo, Mali, and available for the duration of the study.
* For the adult cohort, females of childbearing potential must be willing to use reliable contraception from 21 days prior to study day 0 through the final study visit as described below.

  * Reliable methods of birth control include 1 of the following: confirmed pharmacologic contraceptives via parenteral delivery or intrauterine or implantable device.
  * Nonchildbearing women will be required to report date of last menstrual period, history of surgical sterility (i.e., tubal ligation, hysterectomy) or premature ovarian insufficiency, and will have urine or serum pregnancy test performed per protocol.

Year 2 Extension Inclusion Criteria:

* Participated in the first year of the protocol.
* Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
* In good general health and without clinically significant medical history.
* Parent and/or guardian able to provide informed consent.
* Willing to have blood samples and data stored for future research.
* Resides in or near Kalifabougou or Torodo, Mali, and available for the duration of the study.

Exclusion Criteria:

* Body weight <15 kg or >30 kg for children, or >60 kg for adults.
* Currently receiving or planning to receive seasonal malaria chemoprevention (SMC).
* Any history of menses (for 6-10 year old cohort) or positive pregnancy test at screening (for adult cohort).
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and comply with the study protocol.
* Subject (for adult subjects) or parental (for minor subjects) study comprehension examination score of <80% correct or per investigator discretion.
* Hemoglobin, white blood cell, absolute neutrophil, or platelet count outside the local laboratory-defined limits of normal. (Subjects may be included at the investigator's discretion for "not clinically significant" values.)
* Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratory-defined upper limit of normal. (Subjects may be included at the investigator's discretion for "not clinically significant" values.)
* Infected with HIV, hepatitis C virus (HCV), or hepatitis B virus (HBV).
* Known or documented sickle cell disease by history. (Note: Known sickle cell trait is NOT exclusionary.)
* Clinically significant abnormal electrocardiogram (ECG; Corrected QT Interval (QTc) >460 or other significant abnormal findings, including unexplained tachycardia or bradycardia).
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.
* Receipt of any investigational product within the past 30 days.
* Participation or planned participation in an interventional trial with an investigational product before the last required protocol visit. (Note: Past, current, or planned participation in observational studies is NOT exclusionary.)
* Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* History of a severe allergic reaction or anaphylaxis.
* Severe asthma (defined as asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past 2 years, or that has required the use of oral or parenteral corticosteroids at any time during the past 2 years).
* Salivary gland disorder diagnosed by a doctor (e.g., parotitis, sialadenitis, sialolithiasis, salivary gland tumors).
* Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, or autoimmune thrombocytopenia.
* Known immunodeficiency syndrome.
* Known asplenia or functional asplenia.
* Use of chronic (≥14 days) oral or IV corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/day) or immunosuppressive drugs within 30 days of day 0.
* Receipt of a live vaccine within the past 4 weeks or a killed vaccine or COVID-19 vaccine within the past 2 weeks prior to study agent administration.
* Receipt of immunoglobulins and/or blood products within the past 6 months.
* Previous receipt of an investigational malaria vaccine or monoclonal antibody in the last 5 years.
* Known allergies or contraindication against artemether-lumefantrine.
* Clinical signs of malnutrition.
* Other condition(s) that, in the opinion of the investigator, would jeopardize the safety or rights of a subject participating in the trial, interfere with the evaluation of the study objectives, or render the subject unable to comply with the protocol.

Year 2 Extension Exclusion Criteria:

* Currently receiving or planning to receive SMC.
* Any history of menses.
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and comply with the study protocol.
* Parental study comprehension examination score of <80% correct or per investigator discretion.
* Hemoglobin, white blood cell, absolute neutrophil, or platelet count outside the local laboratory-defined limits of normal. (Subjects may be included at the investigator's discretion for "not clinically significant" values.)
* Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratory-defined upper limit of normal. (Subjects may be included at the investigator's discretion for "not clinically significant" values.)
* Infected with HIV, hepatitis C virus (HCV), or hepatitis B virus (HBV).
* Known or documented sickle cell disease by history. (Note: Known sickle cell trait is NOT exclusionary.)
* Clinically significant abnormal electrocardiogram (ECG; QTc >460 or other significant abnormal findings, including unexplained tachycardia or bradycardia).
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.
* Receipt of any investigational product within the past 30 days.
* Participation or planned participation in another interventional trial with an investigational product other than L9LS until the last required protocol visit. (Note: Past, current, or planned participation in observational studies is NOT exclusionary.)
* Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* History of a severe allergic reaction or anaphylaxis.
* Severe asthma (defined as asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past 2 years, or that has required the use of oral or parenteral corticosteroids at any time during the past 2 years).
* Currently active salivary gland disorder diagnosed by a doctor (e.g., parotitis, sialadenitis, sialolithiasis, salivary gland tumors).
* Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, or autoimmune thrombocytopenia.
* Known immunodeficiency syndrome.
* Known asplenia or functional asplenia.
* Use of chronic (≥14 days) oral or IV corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/day) or immunosuppressive drugs within 30 days of day 0.
* Receipt of a live vaccine within the past 4 weeks or a killed vaccine or COVID-19 vaccine within the past 2 weeks prior to study agent administration.
* Receipt of immunoglobulins and/or blood products within the past 6 months.
* Previous receipt of an investigational malaria vaccine or any other monoclonal antibody other than L9LS in the last 5 years.
* Known allergies or contraindication against artemether-lumefantrine.
* Clinical signs of malnutrition.
* Other condition(s) that, in the opinion of the investigator, would jeopardize the safety or rights of a subject participating in the trial, interfere with the evaluation of the study objectives, or render the subject unable to comply with the protocol.

Ages: 6 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 365 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kassoum Kayentao, MD, MPH, PhD, Principal Investigator — Faculté de Médecine Pharmacie d'Odontostomatologie (FMPOS); Peter Crompton, MD, MPH, Principal Investigator — National Institutes of Health (NIH)
Locations (2):
- Mali (2):
  - Kalifabougou MRTC Clinic, Kalifabougou, Koulikoro
  - Torodo MRTC Clinic, Torodo, Koulikoro

IPD SHARING:
Plan to Share IPD: Yes
Human data generated in this study for future research will be shared as follows:
  * De-identified or identified data with approved outside collaborators under appropriate agreements.
  * De-identified results or data in publication and/or public presentations.
Supporting Information: Study Protocol
Time Frame: Data will be shared at the time of publication or shortly thereafter.
Access Criteria: Data from this study may be requested from other researchers indefinitely after the completion of the primary endpoint by contacting Laboratory of Immunogenetics at NIH

REFERENCES:
- [Result] Kayentao K, Ongoiba A, Preston AC, Healy SA, Hu Z, Skinner J, Doumbo S, Wang J, Cisse H, Doumtabe D, Traore A, Traore H, Djiguiba A, Li S, Peterson ME, Telscher S, Idris AH, Adams WC, McDermott AB, Narpala S, Lin BC, Serebryannyy L, Hickman SP, McDougal AJ, Vazquez S, Reiber M, Stein JA, Gall JG, Carlton K, Schwabl P, Traore S, Keita M, Zeguime A, Ouattara A, Doucoure M, Dolo A, Murphy SC, Neafsey DE, Portugal S, Djimde A, Traore B, Seder RA, Crompton PD; Mali Malaria mAb Trial Team. Subcutaneous Administration of a Monoclonal Antibody to Prevent Malaria. N Engl J Med. 2024 May 2;390(17):1549-1559. doi: 10.1056/NEJMoa2312775. Epub 2024 Apr 26. PMID 38669354

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 365 participants were consented (341 pediatrics, 36 adults):
  * 62 participants were ineligible (57 pediatrics, five adults)
  * 23 participants served as backup (22 pediatrics, one adult)
  * One pediatric participant withdrew consent
  * 279 participants received intervention (261 pediatrics, 18 adults) in year one
  * 235 pediatric participants from year one participated in the extension study in year two
Groups:
- Adult Dose-escalation Study: Arm 1: 300 mg of L9LS: Adult participants receive single dose of 300 mg of L9LS subcutaneously. Once subjects reach day 7 post-administration without safety concerns dosing begins for arm 2.
  L9LS (VRC-MALMAB0114-00-AB): Administered one time via subcutaneous route.
- Adult Dose-escalation Study: Arm 2: 600 mg of L9LS: Adult participants receive single dose of 600 mg of L9LS subcutaneously. Once subjects reach day 7 post-administration without safety concerns dosing begins for arm 3.
  L9LS (VRC-MALMAB0114-00-AB): Administered one time via subcutaneous route.
- Adult Dose-escalation Study: Arm 3: 20 mg/kg of L9LS: Adult participants receive highest single dose of 20 mg/kg IV of L9LS intravenously. Once subjects reach day 7 post-administration without safety concerns dosing begins for pediatric subjects dose escalation arm 1.
  L9LS (VRC-MALMAB0114-00-AB): Administered one time via intravenous route.
- Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS: Pediatric subjects ages 6-10 years receive 150 mg of L9LS subcutaneously. Once subjects reach day 7 post-administration without safety concerns, dosing begins for arm 2.
  L9LS (VRC-MALMAB0114-00-AB): Administered one time via subcutaneous route.
- Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS: Pediatric subjects ages 6-10 years receive 300 mg of L9LS subcutaneously. Once subjects reach day 7 post-administration without safety concerns, dosing begins for the pediatric efficacy study arms.
  L9LS (VRC-MALMAB0114-00-AB): Administered one time via subcutaneous route.
- Pediatric Dose-escalation Study: Arm 3: Placebo; Pediatric Efficacy Study: Arm 3: Placebo: Pediatric subjects ages 6-10 receive placebo of normal saline subcutaneously.
  Normal saline: Administered one time via subcutaneous administration.
- Pediatric Efficacy Study: Arm 1: 150 mg of L9LS: Pediatric subjects ages 6-10 receive 150 mg of L9LS subcutaneously.
  L9LS (VRC-MALMAB0114-00-AB): Administered one time via subcutaneous route.
- Pediatric Efficacy Study: Arm 2: 300 mg of L9LS: Pediatric subjects ages 6-10 receive 300 mg of L9LS subcutaneously.
  L9LS (VRC-MALMAB0114-00-AB): Administered one time via subcutaneous route.
Period: Adult Dose-escalation: 300 mg L9LS
Arm/Group | Adult Dose-escalation Study: Arm 1: 300 mg of L9LS | Adult Dose-escalation Study: Arm 2: 600 mg of L9LS | Adult Dose-escalation Study: Arm 3: 20 mg/kg of L9LS | Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS | Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS | Pediatric Dose-escalation Study: Arm 3: Placebo | Pediatric Efficacy Study: Arm 1: 150 mg of L9LS | Pediatric Efficacy Study: Arm 2: 300 mg of L9LS | Pediatric Efficacy Study: Arm 3: Placebo | Pediatric Extension Study: Arm 1: 150 mg of L9LS | Pediatric Extension Study: Arm 2: 300 mg of L9LS | Pediatric Extension Study: Arm 3: Placebo
Started | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Adult Dose-escalation: 600 mg L9LS
Arm/Group | Adult Dose-escalation Study: Arm 1: 300 mg of L9LS | Adult Dose-escalation Study: Arm 2: 600 mg of L9LS | Adult Dose-escalation Study: Arm 3: 20 mg/kg of L9LS | Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS | Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS | Pediatric Dose-escalation Study: Arm 3: Placebo | Pediatric Efficacy Study: Arm 1: 150 mg of L9LS | Pediatric Efficacy Study: Arm 2: 300 mg of L9LS | Pediatric Efficacy Study: Arm 3: Placebo | Pediatric Extension Study: Arm 1: 150 mg of L9LS | Pediatric Extension Study: Arm 2: 300 mg of L9LS | Pediatric Extension Study: Arm 3: Placebo
Started | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Adult Dose-escalation: 20 mg/kg L9LS
Arm/Group | Adult Dose-escalation Study: Arm 1: 300 mg of L9LS | Adult Dose-escalation Study: Arm 2: 600 mg of L9LS | Adult Dose-escalation Study: Arm 3: 20 mg/kg of L9LS | Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS | Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS | Pediatric Dose-escalation Study: Arm 3: Placebo | Pediatric Efficacy Study: Arm 1: 150 mg of L9LS | Pediatric Efficacy Study: Arm 2: 300 mg of L9LS | Pediatric Efficacy Study: Arm 3: Placebo | Pediatric Extension Study: Arm 1: 150 mg of L9LS | Pediatric Extension Study: Arm 2: 300 mg of L9LS | Pediatric Extension Study: Arm 3: Placebo
Started | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Ped Dose-escalation: 150mg L9LS/ Placebo
Arm/Group | Adult Dose-escalation Study: Arm 1: 300 mg of L9LS | Adult Dose-escalation Study: Arm 2: 600 mg of L9LS | Adult Dose-escalation Study: Arm 3: 20 mg/kg of L9LS | Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS | Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS | Pediatric Dose-escalation Study: Arm 3: Placebo | Pediatric Efficacy Study: Arm 1: 150 mg of L9LS | Pediatric Efficacy Study: Arm 2: 300 mg of L9LS | Pediatric Efficacy Study: Arm 3: Placebo | Pediatric Extension Study: Arm 1: 150 mg of L9LS | Pediatric Extension Study: Arm 2: 300 mg of L9LS | Pediatric Extension Study: Arm 3: Placebo
Started | 0 | 0 | 0 | 9 | 0 | 9 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 9 | 0 | 9 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Ped Dose-escalation: 300mg L9LS/ Placebo
Arm/Group | Adult Dose-escalation Study: Arm 1: 300 mg of L9LS | Adult Dose-escalation Study: Arm 2: 600 mg of L9LS | Adult Dose-escalation Study: Arm 3: 20 mg/kg of L9LS | Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS | Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS | Pediatric Dose-escalation Study: Arm 3: Placebo | Pediatric Efficacy Study: Arm 1: 150 mg of L9LS | Pediatric Efficacy Study: Arm 2: 300 mg of L9LS | Pediatric Efficacy Study: Arm 3: Placebo | Pediatric Extension Study: Arm 1: 150 mg of L9LS | Pediatric Extension Study: Arm 2: 300 mg of L9LS | Pediatric Extension Study: Arm 3: Placebo
Started | 0 | 0 | 0 | 0 | 9 | 9 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 9 | 9 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Pediatric Efficacy Study
Arm/Group | Adult Dose-escalation Study: Arm 1: 300 mg of L9LS | Adult Dose-escalation Study: Arm 2: 600 mg of L9LS | Adult Dose-escalation Study: Arm 3: 20 mg/kg of L9LS | Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS | Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS | Pediatric Dose-escalation Study: Arm 3: Placebo | Pediatric Efficacy Study: Arm 1: 150 mg of L9LS | Pediatric Efficacy Study: Arm 2: 300 mg of L9LS | Pediatric Efficacy Study: Arm 3: Placebo | Pediatric Extension Study: Arm 1: 150 mg of L9LS | Pediatric Extension Study: Arm 2: 300 mg of L9LS | Pediatric Extension Study: Arm 3: Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 75 | 75 | 75 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 73 | 74 | 72 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrew consent | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Period: Pediatric Extension Study
Arm/Group | Adult Dose-escalation Study: Arm 1: 300 mg of L9LS | Adult Dose-escalation Study: Arm 2: 600 mg of L9LS | Adult Dose-escalation Study: Arm 3: 20 mg/kg of L9LS | Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS | Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS | Pediatric Dose-escalation Study: Arm 3: Placebo | Pediatric Efficacy Study: Arm 1: 150 mg of L9LS | Pediatric Efficacy Study: Arm 2: 300 mg of L9LS | Pediatric Efficacy Study: Arm 3: Placebo | Pediatric Extension Study: Arm 1: 150 mg of L9LS | Pediatric Extension Study: Arm 2: 300 mg of L9LS | Pediatric Extension Study: Arm 3: Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 79 | 38 | 118
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 79 | 37 | 116
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adult Dose-escalation Study: Arm 1: 300 mg of L9LS | Adult Dose-escalation Study: Arm 2: 600 mg of L9LS | Adult Dose-escalation Study: Arm 3: 20 mg/kg of L9LS | Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS | Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS | Pediatric Dose-escalation Study: Arm 3: Placebo | Pediatric Efficacy Study: Arm 1: 150 mg of L9LS | Pediatric Efficacy Study: Arm 2: 300 mg of L9LS | Pediatric Efficacy Study: Arm 3: Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 9 | 9 | 18 | 75 | 75 | 75 | 279
Age, Customized [Count of Participants; unit: Participants]
  6 | 0 | 0 | 0 | 0 | 1 | 5 | 20 | 23 | 31 | 80
  7 | 0 | 0 | 0 | 3 | 2 | 4 | 11 | 11 | 8 | 39
  8 | 0 | 0 | 0 | 3 | 2 | 4 | 23 | 13 | 19 | 64
  9 | 0 | 0 | 0 | 1 | 3 | 2 | 15 | 15 | 9 | 45
  10 | 0 | 0 | 0 | 2 | 1 | 3 | 6 | 13 | 8 | 33
  18-20 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  21-30 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  31-40 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  41-50 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  51-55 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 7 | 3 | 8 | 31 | 33 | 36 | 129
  Male | 3 | 2 | 2 | 2 | 6 | 10 | 44 | 42 | 39 | 150
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African | 6 | 6 | 6 | 9 | 9 | 18 | 75 | 75 | 75 | 279
Region of Enrollment [Number; unit: participants]
  Mali | 6 | 6 | 6 | 9 | 9 | 18 | 75 | 75 | 75 | 279

OUTCOME MEASURES:

1. Primary Outcome: Participants With Local Adverse Events (AEs) - Year One
Description: Number of participants with local adverse events occurring within 7 days after administration of L9LS. Local reactogenicity included pain/tenderness, swelling, redness, bruising, and pruritus at the site of infusion. Adverse events were captured by Investigator examination and history from participants.
Time Frame: Within 7 days after administration of L9LS
Population: Modified intention-to-treat (MITT) - Analysis include all randomized subjects that received the study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS: Pediatric subjects age 6-10 years receive 150 mg of L9LS subcutaneously. Once subjects reach day 7 post-administration without safety concerns, dosing begins for arm 2.
  L9LS (VRC-MALMAB0114-00-AB): Administered one time via subcutaneous route.
- Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS: Pediatric subjects age 6-10 years receive 300 mg of L9LS subcutaneously. Once subjects reach day 7 post-administration without safety concerns, dosing begins for the pediatric efficacy study arms.
  L9LS (VRC-MALMAB0114-00-AB): Administered one time via subcutaneous route.
- Pediatric Dose-escalation Study: Arm 3: Placebo; Pediatric Efficacy Study: Arm 3: Placebo: Pediatric subjects age 6-10 receive placebo of normal saline subcutaneously.
  Normal saline: Administered one time via subcutaneous administration.
- Pediatric Efficacy Study: Arm 1: 150 mg of L9LS: Pediatric subjects age 6-10 receive 150 mg of L9LS subcutaneously.
  L9LS (VRC-MALMAB0114-00-AB): Administered one time via subcutaneous route.
- Pediatric Efficacy Study: Arm 2: 300 mg of L9LS: Pediatric subjects age 6-10 receive 300 mg of L9LS subcutaneously.
  L9LS (VRC-MALMAB0114-00-AB): Administered one time via subcutaneous route.
Arm/Group | Adult Dose-escalation Study: Arm 1: 300 mg of L9LS | Adult Dose-escalation Study: Arm 2: 600 mg of L9LS | Adult Dose-escalation Study: Arm 3: 20 mg/kg of L9LS | Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS | Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS | Pediatric Dose-escalation Study: Arm 3: Placebo | Pediatric Efficacy Study: Arm 1: 150 mg of L9LS | Pediatric Efficacy Study: Arm 2: 300 mg of L9LS | Pediatric Efficacy Study: Arm 3: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 9 | 9 | 18 | 75 | 75 | 75
Participants
  Injection site swelling | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0
  Pain at Injection site | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Tenderness at injection site | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness at injection site | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bruising at injection site | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pruritus at injection site | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Severity of Local Adverse Events (AEs) - Year One
Description: The severity of local AEs was graded using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Clinical Trials.
  Grade 1: Pain = does not interfere with activity; Tenderness = mild discomfort to touch; Erythema/Redness = 2.5-5 cm; Induration/Swelling = 2.5-5 cm and does not interfere with activity.
  Grade 2: Pain = Repeated use of non-narcotic pain reliever > 24 hours or interferes with daily activity; Tenderness= Discomfort with movement; Erythema/Redness = 5.1-10 cm; Induration/Swelling = 5.1-10 cm and interferes with activity.
  Grade 3: Pain = Any use of narcotic pain reliever or prevents daily activity; Tenderness = Significant discomfort at rest; Erythema/Redness = > 10 cm; Induration/Swelling = > 10 cm or prevents daily activity.
  Grade 4: Pain = Emergency room (ER) visit or hospitalization; Tenderness = ER visit or hospitalization; Erythema/Redness = Necrosis or exfoliative dermatitis; induration/Swelling = Necrosis
  Grade 5: Death
Time Frame: Within 7 days after administration of L9LS
Population: Modified intention-to-treat (MITT) - Analysis include all randomized subjects that received the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Dose-escalation Study: Arm 1: 300 mg of L9LS | Adult Dose-escalation Study: Arm 2: 600 mg of L9LS | Adult Dose-escalation Study: Arm 3: 20 mg/kg of L9LS | Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS | Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS | Pediatric Dose-escalation Study: Arm 3: Placebo | Pediatric Efficacy Study: Arm 1: 150 mg of L9LS | Pediatric Efficacy Study: Arm 2: 300 mg of L9LS | Pediatric Efficacy Study: Arm 3: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 9 | 9 | 18 | 75 | 75 | 75
Participants
  Grade 1 | 3 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 2
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Participants With Systemic Adverse Events (AEs) - Year One
Description: Number of participants with local adverse events occurring within 7 days after administration of L9LS. Systemic reactogenicity events included fever, feeling unusually tired or unwell, muscle aches, headache, chills, nausea, and joint pain. Adverse events were captured by Investigator examination and history from participants.
Time Frame: Within 7 days after the administration of L9LS
Population: Modified intention-to-treat (MITT) - Analysis include all randomized subjects that received the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Dose-escalation Study: Arm 1: 300 mg of L9LS | Adult Dose-escalation Study: Arm 2: 600 mg of L9LS | Adult Dose-escalation Study: Arm 3: 20 mg/kg of L9LS | Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS | Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS | Pediatric Dose-escalation Study: Arm 3: Placebo | Pediatric Efficacy Study: Arm 1: 150 mg of L9LS | Pediatric Efficacy Study: Arm 2: 300 mg of L9LS | Pediatric Efficacy Study: Arm 3: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 9 | 9 | 18 | 75 | 75 | 75
Participants
  Fever | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1
  Feeling unusually tired or unwell | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Muscle aches | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1
  Chills | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Nausea | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Joint pain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Severity of Systemic Adverse Events (AEs) - Year One
Description: The severity of systemic AEs occurring after the administration of L9LS was assessed using the grading scale below:
  Grade 1: Fever = 37.5^oC-37.9^oC; Fatigue, Headache, Myalgia = No interference with activity; Nausea = no interference with activity or 1-2 episodes/hour
  Grade 2: Fever = 38^oC-38.4^oC; Fatigue, Myalgia = Some interference with activity; Headache = Repeated use of non-narcotic pain reliever > 24 hours or some interference with activity; Nausea = Some interference with activity or > 2 episodes/24 hours
  Grade 3: Fever = 38.5^oC-39.5^oC; Fatigue = Prevents daily activity; Headache =Significant; any use of narcotic pain reliever or prevents daily activity; Myalgia =Significant; prevents daily activity; Nausea = Prevents daily activity, requires outpatient intravenous hydration
  Grade 4: Fever = > 39.5^oC; Fatigue, Headache, Myalgia = Emergency room (ER) visit or hospitalization; Nausea = ER visit or hospitalization for hypotensive shock
  Grade 5: Death
Time Frame: Within 7 days after the administration of L9LS
Population: Modified intention-to-treat (MITT) - Analysis include all randomized subjects that received the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Dose-escalation Study: Arm 1: 300 mg of L9LS | Adult Dose-escalation Study: Arm 2: 600 mg of L9LS | Adult Dose-escalation Study: Arm 3: 20 mg/kg of L9LS | Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS | Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS | Pediatric Dose-escalation Study: Arm 3: Placebo | Pediatric Efficacy Study: Arm 1: 150 mg of L9LS | Pediatric Efficacy Study: Arm 2: 300 mg of L9LS | Pediatric Efficacy Study: Arm 3: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 9 | 9 | 18 | 75 | 75 | 75
Participants
  Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Participants With Plasmodium Falciparum (Pf) Infection Detected by Microscopic Examination - Efficacy Study
Description: Number of participants with Plasmodium falciparum (Pf) blood stage infection defined as blood smear-positive for Pf was assessed by microscopic examination of thick blood smear collected from participants from day 14 through week 28 (196 days) after administration of L9LS or placebo. Analysis was done as number of participants who had at least one positive blood smear.
Time Frame: Day 7 through week 28
Population: Modified intention-to-treat (MITT) - Analysis include all randomized subjects that received the study intervention during the efficacy study.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Efficacy Study: Arm 1: 150 mg of L9LS | Pediatric Efficacy Study: Arm 2: 300 mg of L9LS | Pediatric Efficacy Study: Arm 3: Placebo
Number analyzed (Participants) | 75 | 75 | 75
Participants | 36 | 30 | 61

6. Primary Outcome: Participants With Detectable Anti-drug Antibody (ADA) in Sera - Extension Study
Description: Number of participants with detectable anti-drug antibody (ADA) in sera after exposure to L9LS. Serum was collected from participants at specific timepoints throughout the study, on days 0, 7, 28, 84, 168, and 196. The tier 3 assay was used to directly measure ADA's ability to impair L9LS binding to Plasmodium falciparum circumsporozoite protein (PfCSP). Analysis was done to determine number of participants with positive or detectable ADA in sera.
Time Frame: Measured through week 36
Population: Modified intention-to-treat (MITT) - Analysis include all randomized subjects that received the study intervention in the extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Extension Study: Arm 1: 150 mg of L9LS | Pediatric Extension Study: Arm 2: 300 mg of L9LS | Pediatric Extension Study: Arm 3: Placebo
Number analyzed (Participants) | 79 | 38 | 118
Participants | 0 | 0 | 0

7. Primary Outcome: Maximum Total Plasma Concentration (Cmax) for L9LS - Extension Study
Description: Maximum total plasma concentration (Cmax) following a dose of 150 mg or 300 mg L9LS. Serum collected on days 0, 7, 28, 84, 140, 196, & 252 after the administration of L9LS. Cmax for L9LS was obtained directly by visual inspection of the plasma concentration versus time profiles post dose. Analysis was done to determine each participant's observed maximum concentration based on all available timepoints and cumulative output was calculated as the central tendency and dispersion metric based on the observed maximum concentrations.
Time Frame: Measured through Week 36
Population: Modified intention-to-treat (MITT) - Analysis include all randomized subjects that received the L9LS intervention during the extension study.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Pediatric Extension Study: Arm 1: 150 mg of L9LS | Pediatric Extension Study: Arm 2: 300 mg of L9LS
Number analyzed (Participants) | 79 | 38
ug/mL | 64.63 (17.36) | 116.93 (24.78)

8. Primary Outcome: Time to Maximum Plasma Concentration (TMax) for L9LS - Extension Study
Description: Time to maximum total plasma concentration (Cmax) following a dose of 150 mg or 300 mg L9LS. Serum collected on days 0, 7, 28, 84, 140, 196, & 252 after the administration of L9LS. Tmax for L9LS was obtained directly by visual inspection of the plasma concentration versus time profiles. Analysis was done to determine the time (in days) at which the maximum observed concentration was achieved for each participant and cumulative output was calculated as the central tendency and dispersion metric based on the observed time of maximum concentration.
Time Frame: Measured through Week 36
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Pediatric Extension Study: Arm 1: 150 mg of L9LS | Pediatric Extension Study: Arm 2: 300 mg of L9LS
Number analyzed (Participants) | 79 | 38
Days | 7.00 (0.16) | 7.58 (3.41)

9. Primary Outcome: Participants With Local Adverse Events (AEs) - Extension Study
Description: as for outcome 1
Time Frame: Within 7 days after administration of L9LS
Population: Modified intention-to-treat (MITT) - Analysis include all randomized subjects that received the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Extension Study: Arm 1: 150 mg of L9LS | Pediatric Extension Study: Arm 2: 300 mg of L9LS | Pediatric Extension Study: Arm 3: Placebo
Number analyzed (Participants) | 79 | 38 | 118
Participants
  Injection site swelling | 1 | 2 | 0
  Pain at Injection site | 0 | 0 | 1
  Tenderness at injection site | 0 | 0 | 0
  Redness at injection site | 0 | 0 | 0
  Bruising at injection site | 0 | 0 | 0
  Pruritus at injection site | 0 | 0 | 0

10. Primary Outcome: Severity of Local Adverse Events (AEs) - Extension Study
Description: as for outcome 2
Time Frame: Within 7 days after administration of L9LS
Population: Modified intention-to-treat (MITT) - Analysis include all randomized subjects that received the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Extension Study: Arm 1: 150 mg of L9LS | Pediatric Extension Study: Arm 2: 300 mg of L9LS | Pediatric Extension Study: Arm 3: Placebo
Number analyzed (Participants) | 79 | 38 | 118
Participants
  Grade 1 | 1 | 2 | 1
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

11. Primary Outcome: Participants With Systemic Adverse Events (AEs) - Extension Study
Description: as for outcome 3
Time Frame: Within 7 days after the administration of L9LS
Population: Modified intention-to-treat (MITT) - Analysis include all randomized subjects that received the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Extension Study: Arm 1: 150 mg of L9LS | Pediatric Extension Study: Arm 2: 300 mg of L9LS | Pediatric Extension Study: Arm 3: Placebo
Number analyzed (Participants) | 79 | 38 | 118
Participants
  Fever | 0 | 0 | 0
  Feeling unusually tired or unwell | 0 | 0 | 0
  Muscle aches | 0 | 0 | 0
  Headache | 1 | 1 | 4
  Chills | 0 | 0 | 0
  Nausea | 0 | 0 | 0
  Joint pain | 0 | 0 | 0

12. Primary Outcome: Severity of Systemic Adverse Events (AEs) - Extension Study
Description: as for outcome 4
Time Frame: Within 7 days after the administration of L9LS
Population: Modified intention-to-treat (MITT) - Analysis include all randomized subjects that received the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Extension Study: Arm 1: 150 mg of L9LS | Pediatric Extension Study: Arm 2: 300 mg of L9LS | Pediatric Extension Study: Arm 3: Placebo
Number analyzed (Participants) | 79 | 38 | 118
Participants
  Grade 1 | 0 | 0 | 1
  Grade 2 | 1 | 1 | 3
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

13. Secondary Outcome: Participants With Plasmodium Falciparum (Pf) Infection Detected by Real-Time Polymerase Chain Reaction (RT-PCR)
Description: Number of participants with Plasmodium falciparum (Pf) blood stage infection defined as blood sample positive for Pf was assessed by real-time polymerase chain reaction (RT-PCR) of blood sample collected from participants from day 0 through week 28 (196 days) after administration of L9LS or placebo. Analysis was done as number of participants who had at least one positive blood sample.
Time Frame: Measured through week 24 (dose escalation study) and week 28 (efficacy study)
Population: Modified intention-to-treat (MITT) - Analysis include all randomized pediatric subjects that received intervention during year one of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS | Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS | Pediatric Dose-escalation Study: Arm 3: Placebo | Pediatric Efficacy Study: Arm 1: 150 mg of L9LS | Pediatric Efficacy Study: Arm 2: 300 mg of L9LS | Pediatric Efficacy Study: Arm 3: Placebo
Number analyzed (Participants) | 9 | 9 | 18 | 75 | 75 | 75
Participants | 7 | 8 | 13 | 33 | 32 | 62

14. Secondary Outcome: Participants With Clinical Malaria - Pediatric Dose Escalation Study
Description: Number of pediatric participants with clinical malaria during a single malaria season, defined by an illness accompanied by measured axillary fever ≥37.5°C, or history of fever (subjective or objective) in the previous 24 hours, and Plasmodium falciparum (Pf) asexual parasitemia >5,000 parasites/μL as detected from microscopic examination of thick blood smear. Assessment was done from day 0 through week 28 (196 days) after administration of L9LS or placebo. Subjective data, objective data and blood sample were collected from administration of intervention through week 28. Analysis was done as number of participants who had at least one symptom and positive blood sample.
Time Frame: Measured through Week 28
Population: Modified intention-to-treat (MITT) - Analysis include all randomized subjects that received intervention during the pediatric dose escalation study.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS | Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS | Pediatric Dose-escalation Study: Arm 3: Placebo
Number analyzed (Participants) | 9 | 9 | 18
Participants | 6 | 4 | 11

15. Secondary Outcome: Participants With Clinical Malaria - Pediatric Efficacy Study
Description: as for outcome 14
Time Frame: Measured through Week 28
Population: Modified intention-to-treat (MITT) - Analysis include all randomized subjects that received the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Efficacy Study: Arm 1: 150 mg of L9LS | Pediatric Efficacy Study: Arm 2: 300 mg of L9LS | Pediatric Efficacy Study: Arm 3: Placebo
Number analyzed (Participants) | 75 | 75 | 75
Participants | 21 | 14 | 44

16. Secondary Outcome: Participants With Clinical Malaria Detected by Microscopic Examination of Thick Blood Smear - Pediatric Dose Escalation Study
Description: Number of participants with clinical malaria during a single malaria season, defined by an illness accompanied by any level of Plasmodium Falciparum (Pf) asexual parasitemia as detected from microscopic examination of thick blood smear that results in the administration of anti-malarial treatment.
Time Frame: Measured through Week 28
Population: Modified intention-to-treat (MITT) - Analysis include all randomized subjects that received the intervention during the pediatric dose escalation study.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS | Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS | Pediatric Dose-escalation Study: Arm 3: Placebo
Number analyzed (Participants) | 9 | 9 | 18
Participants | 7 | 7 | 13

17. Secondary Outcome: Participants With Clinical Malaria Detected by Microscopic Examination of Thick Blood Smear - Pediatric Efficacy Study
Description: as for outcome 16
Time Frame: Measured through Week 24
Population: Modified intention-to-treat (MITT) - Analysis include all randomized subjects that received intervention during the pediatric efficacy study.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Efficacy Study: Arm 1: 150 mg of L9LS | Pediatric Efficacy Study: Arm 2: 300 mg of L9LS | Pediatric Efficacy Study: Arm 3: Placebo
Number analyzed (Participants) | 75 | 75 | 75
Participants | 33 | 25 | 57

18. Secondary Outcome: Maximum Total Plasma Concentration (Cmax) for L9LS - Study Year One
Description: Maximum total plasma concentration (Cmax) following a dose of 150 mg or 300 mg L9LS. Serum collected on days 0, 7, 28, 56, 84, 112, 140, 168, 196, 224, & 252 after the administration of L9LS. Cmax for L9LS was obtained directly by visual inspection of the plasma concentration versus time profiles post dose. Analysis was done to determine each participant's observed maximum concentration based on all available timepoints and cumulative output was calculated as the central tendency and dispersion metric based on the observed maximum concentrations.
Time Frame: Measured through Week 36
Population: Modified intention-to-treat (MITT) - Analysis include all randomized subjects that received L9LS in year one study.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS | Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS | Pediatric Efficacy Study: Arm 1: 150 mg of L9LS | Pediatric Efficacy Study: Arm 2: 300 mg of L9LS
Number analyzed (Participants) | 9 | 9 | 75 | 75
ug/mL | 76.97 (18.88) | 142.79 (30.36) | 76.19 (22.04) | 142.70 (29.56)

19. Secondary Outcome: Time to Maximum Plasma Concentration (TMax) for L9LS - Study Year One
Description: Time to maximum total plasma concentration (Cmax) following a dose of 150 mg or 300 mg L9LS. Serum was collected on days 0, 7, 28, 56, 84, 112, 140, 168, 196, 224, & 252 after administration of L9LS. Tmax for L9LS was obtained directly by visual inspection of the plasma concentration versus time profiles. Analysis was done to determine the time (in days) at which the maximum observed concentration was achieved for each participant and cumulative output was calculated as the central tendency and dispersion metric based on the observed time of maximum concentration.
Time Frame: Measured through Week 36
Population: Modified intention-to-treat (MITT) - Analysis include all randomized subjects that received L9LS in year one study.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS | Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS | Pediatric Efficacy Study: Arm 1: 150 mg of L9LS | Pediatric Efficacy Study: Arm 2: 300 mg of L9LS
Number analyzed (Participants) | 9 | 9 | 75 | 75
Days | 7.00 (0.00) | 7.00 (0.00) | 7.17 (2.46) | 7.36 (2.45)

ADVERSE EVENTS:
Time Frame: Up to 196 days for adult dose escalation groups and up to 252 days for the pediatric dose escalation groups, post administration of intervention (year one) Up to 168 days for the efficacy groups, post administration of intervention (year one) Up to 252 days for the extension groups, post administration of intervention (year two)
Arm/Group | Adult Dose-escalation Study: Arm 1: 300 mg of L9LS | Adult Dose-escalation Study: Arm 2: 600 mg of L9LS | Adult Dose-escalation Study: Arm 3: 20 mg/kg of L9LS | Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS | Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS | Pediatric Dose-escalation Study: Arm 3: Placebo | Pediatric Efficacy Study: Arm 1: 150 mg of L9LS | Pediatric Efficacy Study: Arm 2: 300 mg of L9LS | Pediatric Efficacy Study: Arm 3: Placebo | Pediatric Extension Study: Arm 1: 150 mg of L9LS | Pediatric Extension Study: Arm 2: 300 mg of L9LS | Pediatric Extension Study: Arm 3: Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/9 | 0/9 | 0/18 | 0/75 | 0/75 | 0/75 | 0/79 | 0/38 | 0/118
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/9 | 0/9 | 0/18 | 0/75 | 0/75 | 0/75 | 0/79 | 0/38 | 0/118
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 6/6 | 9/9 | 8/9 | 18/18 | 67/75 | 71/75 | 72/75 | 74/79 | 33/38 | 111/118
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adult Dose-escalation Study: Arm 1: 300 mg of L9LS (N=6) | Adult Dose-escalation Study: Arm 2: 600 mg of L9LS (N=6) | Adult Dose-escalation Study: Arm 3: 20 mg/kg of L9LS (N=6) | Pediatric Dose-escalation Study: Arm 1: 150 mg of L9LS (N=9) | Pediatric Dose-escalation Study: Arm 2: 300 mg of L9LS (N=9) | Pediatric Dose-escalation Study: Arm 3: Placebo (N=18) | Pediatric Efficacy Study: Arm 1: 150 mg of L9LS (N=75) | Pediatric Efficacy Study: Arm 2: 300 mg of L9LS (N=75) | Pediatric Efficacy Study: Arm 3: Placebo (N=75) | Pediatric Extension Study: Arm 1: 150 mg of L9LS (N=79) | Pediatric Extension Study: Arm 2: 300 mg of L9LS (N=38) | Pediatric Extension Study: Arm 3: Placebo (N=118)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 2 | 0 | 3 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 2 | 0 | 4 | 1 | 3 | 3 | 2 | 0 | 5
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0
Dizziness (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 2 | 1 | 2 | 0 | 0 | 1 | 4 | 6 | 1 | 1 | 3
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 7 | 19 | 13 | 16 | 26 | 9 | 33
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 4 | 2 | 0 | 2
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 6 | 1 | 2
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site swelling (General disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 1 | 2 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 2 | 1 | 1 | 12 | 13 | 7 | 6 | 1 | 11
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 12 | 3 | 20
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2
Malaria (Infections and infestations) | 1 | 2 | 1 | 7 | 7 | 13 | 36 | 33 | 59 | 32 | 15 | 83
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 2 | 0 | 6
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 1 | 5
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Blood Pressure Diastolic Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 5
Blood pressure systolic decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 5 | 4 | 5 | 2 | 1 | 2
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 2 | 1 | 5 | 3 | 8 | 27 | 27 | 21 | 34 | 10 | 52
Urinary tract infection (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 2 | 3 | 13 | 18 | 22 | 17 | 11 | 22
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 4 | 3 | 3 | 19 | 26 | 27 | 17 | 9 | 24
Tonsillitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 7 | 1 | 10
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 4 | 4 | 4 | 6 | 35 | 36 | 33 | 13 | 10 | 24
Paronychia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinea capitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Diastolic hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Dysentery (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Parotitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Salmonellosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5
Schistosomiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Forearm fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4
Furuncle (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT05304611/Prot_SAP_000.pdf